CLINICAL TRIAL: NCT00998595
Title: Es Mejor Saber: A Proactive Approach to Gestational Diabetes Follow Up
Brief Title: Gestational Diabetes Follow Up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Association of American Medical Colleges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MM-1107-09/09 (AAMC-CDC)
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2011-09

CONDITIONS: Diabetes, Gestational; Postpartum Period
Keywords: Diabetes, Gestational; Postpartum Period; Reproductive Health Services; Health Promotion; Health Personnel
MeSH Terms: conditions — Diabetes, Gestational | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promotora (Experimental): This group receives additional education and proactive follow-up by removing barriers to already existing services and reminders by a lay community health workers (Promotora)
  Interventions: Other: Promotora
- Standard of Care (No Intervention): These subjects receive the routine standard of postpartum care

INTERVENTIONS:
Other: Promotora — The Promotora will deliver education regarding postpartum follow-up and steps to take to decrease the risk for developing type 2 diabetes. The Promotora will clarify misperceptions and answer questions related to risk of developing diabetes and contraception. If the subject has barriers to accessing care with transportation or childcare, she will help the subjects to access existing resources. The Promotora will give the subject her contact information and will also contact the subject to remind her of her appointments and reschedule if she missed an appointment.
  Other Names: Community Health Worker; Lay Community Worker
  Arms: Promotora

SUMMARY:
The primary hypothesis underlying this proposal is that the introduction of a Promotora to provide education and proactive follow-up to women with GDM will increase compliance with postpartum glucose tolerance testing. The secondary hypothesis is that the Promotora will improve participation in referral visits for diabetes or preventive care. We will develop the promotora program and begin pilot implementation.

DETAILED DESCRIPTION:
As Los Angeles County + University of Southern California Medical Center (LAC+USC) serves an indigent Latino population at increased risk for developing Type 2 Diabetes Mellitus (T2DM), Gestational Diabetes Mellitus (GDM) complicated 13% of deliveries at LAC+USC between 2006-2007. While over 50% of GDM patients will develop overt diabetes mellitus within a decade of the incident pregnancy, less than half of these patients ever return for even one post-partum follow up visit at this institution (45%). Lifestyle Interventions and medications have been shown to delay or prevent the onset of T2DM. However, prevention is only possible if patients follow-up and individual risk assessment is made. While identifying the 2-hour glucose tolerance test as the appropriate postpartum screening technique for patients with a history of GDM, the Fifth International Workshop-Conference on Gestational Diabetes Mellitus did not identify strategies to improve follow up among this patient population. Promotoras (bi-lingual, bi-cultural lay community health workers representative of the Latino community base) have been successful in improving follow up for other areas of diabetes and women's preventive services but have not been studies in the context of GDM. We will develop the Es Mejor Saber training materials and program and pilot a randomized control trial (RCT),a total 216 subjects completing a GDM affected pregnancy will be randomized on the postpartum ward to the standard-of-care versus proactive follow-up with a Promotora. The Promotora will provide education, address barriers to follow-up, remind subjects of their appointments, and call them to reschedule if they miss appointments. In the first phase of the study, these appointments will include the OGTT and the initial postpartum visit. In the second phase, these visits will include referrals to internal medicine (for those diagnosed with T2DM) or nutrition counseling (for those found not to have diabetes). The primary hypothesis underlying this proposal is that the introduction of a Promotora providing education and pro-active follow-up into postpartum GDM management will result improve post-partum follow-up for screening, treatment, and preventive services when compared with the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes for the first time during the most recent pregnancy
* Completed pregnancy >20 weeks duration
* Has access to a telephone
* Is willing to be contacted by the Promotora
* Is willing to follow-up at LAC+USC for postpartum visit
* Able to give informed consent
* Age ≥18 years
* Residence within 60 miles of LAC+USC
* ON INPATIENT WARD AT LAC+USC AT TIME OF RECRUITMENT

Exclusion Criteria:

* Diagnosis of diabetes prior to most recent pregnancy (pre-gestational diabetes)
* Current ICU admission during delivery hospitalization that would interfere with recruitment and participation in the study
* Currently residing in jail or inpatient psychiatric facility
* Postpartum day #1-2, any Fasting Blood Glucose ≥126mg/dL or random BG≥200mg/dL
* Plans postpartum follow-up at non-participating postpartum clinic location

A Medical Record Abstraction Only Cohort is a third group of patients who live within 60 miles of LAC+USC, plan to obtain postpartum care at LAC+USC, and completed a GDM affected pregnancy but refuse participation or do not qualify based on the following: elevated glucose consistent with diagnosis of T2DM or maintained on insulin postpartum, incarceration or resides in inpatient psychiatric facility, age <18, no telephone, unwilling to be contacted by Promotora, or are unable to consent for participation.This cohort can not be enrolled in the study but data is abstracted from the medical records to compare demographics and follow up in our study to all patients with GDM who deliver at LAC+USC.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
the fraction of each group that participates in postpartum follow up and glucose tolerance testing 4-12 weeks post partum. | 4-12 weeks post partum

SECONDARY OUTCOMES:
the fraction of women in each group that attends a referral visit | within 8 weeks following referral

CONTACTS AND LOCATIONS:
Overall Officials: Penina Segall-Gutierrez, M.D., M.Sc., Principal Investigator — University of Southern California
Locations (1):
- Los Angeles County + University of Southern California Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Zaman A, Ovalle B, Reyes C, Segall-Gutierrez P. Enhanced Participation in Diabetes Screening and Care After Gestational Diabetes Through Community Health Workers: Results from the Es Mejor Saber Randomized Controlled Trial. J Immigr Minor Health. 2024 Feb;26(1):45-53. doi: 10.1007/s10903-023-01547-5. Epub 2023 Oct 25. PMID 37878217